CLINICAL TRIAL: NCT06922084
Title: A Prospective, Randomized, Subject and Vision-assessor Masked, Multicenter Study Comparing Bilateral Clareon PanOptix, Bilateral Clareon PanOptix Pro, and Mixed Clareon PanOptix Pro/Vivity Intraocular Lens Implantation in Cataract Subjects
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Berkeley Eye Center (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 95474481
Record Dates: First submitted 2025-03-28; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Bilateral Clareon PanOptix IOL implantation (Active Comparator)
  Interventions: Device: Clareon PanOptix
- Bilateral Clareon PanOptix Pro IOL implantation (Experimental)
  Interventions: Drug: Clareon PanOptix PRO
- Clareon PanOptix Pro in the non-dominant eye and Clareon Vivity in the dominant eye (Experimental)
  Interventions: Drug: Mix-and-Match PanOptix/Vivity

INTERVENTIONS:
Device: Clareon PanOptix — Bilateral Clareon PanOptix IOL implantation
  Arms: Bilateral Clareon PanOptix IOL implantation
Drug: Clareon PanOptix PRO — Bilateral Clareon PanOptix PRO IOL implantation
  Arms: Bilateral Clareon PanOptix Pro IOL implantation
Drug: Mix-and-Match PanOptix/Vivity — Clareon PanOptix Pro in the non-dominant eye and Clareon Vivity in the dominant eye
  Arms: Clareon PanOptix Pro in the non-dominant eye and Clareon Vivity in the dominant eye

SUMMARY:
Prospective, randomized, multicenter, multi-arm, subject and vision-assessor-masked, two stage study with Stage 1 as a three-arm initial enrollment period, followed by Stage 2 as a head-to-head study refined based on the Stage 1 data.

ELIGIBILITY:
Inclusion Criteria:

* Adult cataract patients aged 40 years and older scheduled for age related cataract surgery in both eyes.
* Ability to understand and sign an ethics committee-approved informed consent form.
* Willingness and ability to attend all scheduled study visits as required by the protocol.
* Postoperative potential visual acuity of 20/25 or better in each eye, as determined by the investigator.
* Preoperative corneal astigmatism that can be corrected with a T3 or T4 toric IOL, or with a spherical IOL and LRIs or AKs resulting in a predicted postoperative astigmatism of less than 0.5 diopters (D).
* Ability to understand and complete questionnaires.

Exclusion Criteria:

* Women who are pregnant, planning to become pregnant during the study, or breastfeeding.
* Ocular conditions that could confound study results, including moderate to severe corneal pathology, irregular astigmatism, moderate to severe dry eye, preexisting retinal diseases such as macular degeneration or diabetic retinopathy.
* Any form of confirmed glaucomatous damage (ie, mild, moderate, or severe glaucoma).
* Participation in another clinical study that could interfere with the results.
* Systemic conditions that may affect healing or visual outcomes (e.g., uncontrolled diabetes mellitus, certain autoimmune disorders).
* Subjects with nystagmus, strabismus, zonular laxity or dehiscence, and pseudoexfoliation.
* Prior ocular surgery (except for uncomplicated cataract surgery in the fellow eye).
* Participants desiring monovision.
* Any active ocular infection or inflammation (except for routine post-operative inflammation in the fellow eye)
* Psychiatric or cognitive disorders that may impair the ability to comply with study procedures or provide accurate self-assessments.
* RMS total higher-order aberrations (HOAs) >0.70 µm or coma >0.40 µm as measured by tomography or topography with a 4 mm pupil setting.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Binocular photopic CDVA (corrected distance visual acuity) | 3 months postoperatively

SECONDARY OUTCOMES:
Binocular photopic DCIVA (distance corrected intermediate visual acuity) and DCNVA (distance corrected near visual acuity) | 3 months postoperatively
Binocular photopic uncorrected visual acuity at distance (UDVA), intermediate (UIVA), and near (UNVA) | 3 months postoperatively
Binocular photopic small letter contrast sensitivity at 66 cm and 100 cm with refractive distance correction (20/32 line) | 3 months postoperatively
Binocular mesopic high contrast distance corrected visual acuity at distance (CDVA), intermediate (DCIVA), and near (DCNVA). | 3 months postoperatively
Binocular photopic distance corrected defocus curve | 3 months postoperatively
  Obtained by varying the vergence of the stimulus from -3.0 D to +1.0 D in steps of 0.5 D with the best correction for distance vision.
Monocular photopic distance corrected defocus curves | 3 months postoperatively
  Obtained by varying the vergence of the stimulus from -3.0 D to +1.0 D in steps of 0.5 D with the best correction for distance vision.
Binocular mesopic distance corrected contrast sensitivity with and without glare (1.5, 3, 6 & 12 cpd) | 3 months postoperatively
Refractive outcomes | 3 months postoperatively
  Mean residual manifest refraction spherical equivalent (MRSE) and residual astigmatism.
Pupil size | 3 months postoperatively
  Under both photopic and mesopic conditions.
Patient-reported outcomes using a questionnaire about visual disturbances (QUVID) | 3 months postoperatively
Patient-reported outcomes using a questionnaire about IOL satisfaction (IOLSAT) | 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Micheletti, MD, Principal Investigator — Berkeley Eye Center
Locations (2):
- United States (2):
  - Shafer Vision Institute, Plymouth Meeting, Pennsylvania
  - Berkeley Eye Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No